CLINICAL TRIAL: NCT05049512
Title: Low Dose Multi-Nut Oral Immunotherapy in Pre-schoolers (LMNOP): a Pragmatic Randomised Controlled Trial of Low Dose Multi-Nut Oral Immunotherapy Versus Standard Care for the Treatment of Multi-Nut Allergies in Young Children
Brief Title: Low Dose Multi-Nut Oral Immunotherapy in Pre-schoolers With a Multi-Nut Allergy
Acronym: LMNOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74540
Record Dates: First submitted 2021-09-08; First posted 2021-09-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Allergy, Nut
Keywords: Oral immunotherapy; Randomised controlled trial; Skin prick test; Oral food challenge
MeSH Terms: conditions — Nut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-nut OIT (Experimental): Participants will have a personalised combination of two nuts they are allergic to for their multi-nut OIT (a. peanut, b. almond, c. cashew, d. hazelnut, e. walnut). In the escalation visit, participants will receive 5 increasing doses of personalised multi-nut OIT in clinic at 20-minute intervals: 1 mg, 3 mg, 6 mg, 12 mg, 24 mg total nut protein, 12 mg/nut. The build-up phase will consist of daily home doses of multi-nut OIT and clinic visits every 2 weeks for up-dosing, up to a maintenance dose of 600 mg total protein, 300 mg/nut, over 3-8 months. In the maintenance phase, participants will continue to take their multi-nut OIT dose of 600 mg total protein each day at home for the remainder of the 18 months, with visits to the clinic every 3 months.
  Interventions: Other: Multi-nut OIT
- Standard Care (No Intervention): Strict avoidance of the 2 study nuts the participants are allergic to over 18 months - a. peanut, b. almond, c. cashew, d. hazelnut, e. walnut, as per standard care instructions for children with allergies in Australia.

INTERVENTIONS:
Other: Multi-nut OIT — Finely ground pure peanut, almond, cashew, hazelnut, and walnut.
  Arms: Multi-nut OIT

SUMMARY:
The LMNOP trial will be a 2-armed, open-label, randomised controlled trial (RCT), 2:1. Over a period of 18 months, children in the Multi-Nut Oral Immunotherapy Treatment (OIT) Group (experimental arm) will undergo low dose OIT to two nuts they are allergic to. At this time, children in the Standard Care Group (control arm) will be instructed to strictly avoid consuming two nuts they are allergic to. Avoiding consuming nut allergens is the standard care advice for children with peanut/tree nut allergies in Australia. The trial will assess the difference in the proportion of participants undergoing Multi-Nut OIT who can achieve sustained unresponsiveness (SU) compared to the proportion of participants avoiding nuts who develop natural tolerance (NT), i.e. grow out of their allergy. SU is when a participant can pass an oral food challenge (OFC) after having paused OIT treatment for several weeks. Participants will be between the ages of 18 and 36 months at the time of screening. The first 12 participants enrolled will be part of the pilot phase, with a total of n = 45 for the main trial.

It is hypothesised that there will be a higher proportion of participants in the Multi-Nut OIT Group versus the Standard Care Group who pass the OFC following the 18-month treatment phase. That is, a higher proportion of participants in the Multi-Nut OIT Group will achieve SU compared to participants in the Standard Care Group achieving NT.

DETAILED DESCRIPTION:
The LMNOP trial is a novel RCT assessing whether, over a period of 18 months, children undergoing low dose, multi-nut OIT can safely achieve SU at a higher rate than children under standard care who develop NT to peanut and tree nuts.

Trial Time Line

Study Entry - Children will undergo a screening skin prick test (SPT) to two of peanut, cashew, almond, hazelnut and/or walnut and OFC.

Children who meet the study eligibility criteria will be randomisation to either the Multi-Nut OIT Group or Standard Care Group for 18 months.

Multi-Nut OIT Group:

The 18-month treatment phase involves an escalation visit, build-up phase and maintenance phase. In the escalation visit, participants will receive 5 increasing doses of personalised multi-nut OIT in clinic at 20-minute intervals: 1 mg, 3 mg, 6 mg, 12 mg, 24 mg total nut protein, 12 mg/nut. The build-up phase will consist of daily home doses of multi-nut OIT and clinic visits every 2 weeks for up-dosing, up to a maintenance dose of 600 mg total protein, 300 mg/nut, over 3-8 months. In the maintenance phase, participants will continue to take their multi-nut OIT dose of 600 mg total protein each day at home for the remainder of the 18 months, with visits to the clinic every 3 months. 300 mg per allergen was chosen as the daily maintenance dose, as this is the lowest dose thus far demonstrated in any trial to successfully achieve SU.

Each dose will be mixed into a carrier food of the participant's choice (e.g. apple puree, custard, chocolate pudding etc).

At the end of the 18-month treatment phase, participants will have a SPT and OFC to their study nuts.

Participants who pass the OFC will cease OIT for 4 weeks. They will then undergo another OFC, 19 months after commencing treatment. Participants who pass this OFC will then enter the Ad libitum phase for 12 months. The Ad libitum phase involves participants eating the study nuts as much or as often as they want. To ensure the participant is consuming some nuts, they will be given advice that at a minimum, participants should have approximately ½ -1 teaspoon of nut flour, twice per week, for each nut.

At the end of the Ad libitum phase, participants will undergo another OFC.

Standard Care Group:

At the end of the 18-month period, participants will have a SPT and OFC to their study nuts.

Participants who pass their OFC will enter Ad libitum Phase for 12 months. As described for the Multi-Nut OIT Group, this involves participants eating the study nuts as much or as often as they want, with advice given that participants should have approximately ½ -1 teaspoon of nut flour, twice per week for each nut at a minimum.

At the end of the Ad libitum phase, participants will undergo another OFC.

Any Multi-Nut OIT Group participants who fail their OFC to one or both of their study nuts after the 18-month treatment phase will be asked to cease OIT to that nut(s) and will be referred back to their regular allergist. Likewise, any Multi-Nut OIT Group participants who fail their OFC to one or both of their study nuts after the 4 weeks of ceasing OIT will be asked to avoid the nut/s and will be referred back to their regular allergist. Any Standard Care Group participants who fail their OFC at this time, will be asked to continue avoiding that nut(s) and will also be referred back to their regular allergist. Participants in both groups who fail their OFC to both study nuts will be invited back at the end of the trial for a clinical assessment, but no OFC.

Primary Aim of the Pilot Phase:

To determine the feasibility of this study design in terms of recruitment into the study and completion of the escalation and build-up phases for participants in the Multi-Nut OIT Group.

Primary Aim of the Main Trial:

To compare the proportion of participants in the Multi-Nut OIT Group versus the Standard Care Group who pass the OFC after the 18-month treatment phase. That is, comparing the proportion of participants in the Multi-Nut OIT Group who achieve SU by passing their OFC after 18 months of OIT, and then passing another OFC after 4 weeks of ceasing OIT, to participants in the Standard Care Group who achieve NT by passing their OFC after the 18-month period.

Healthy children aged 18-36 months at the screening visit with confirmed/suspected Immunoglobulin E-mediated (IgE-mediated) allergies to 2 of: peanut, cashew, almond, hazelnut and/or walnut, and who meet the study criteria, will be recruited into the trial. Children will be randomised (2:1) for the pilot phase to either: multi-nut OIT (n ~ 8) or standard care (n ~ 4), and for the main trial - multi-nut OIT (n ~ 30) or standard care (n ~ 15). The 12 pilot participants will be included in the over all total of 45 participants.

Data from the first 12 participants enrolled, denoted the Pilot Phase, will be used to assess the feasibility of our study design in terms of the screening, recruitment, randomisation and treatment of participants, and examine the acceptability of low dose, multi-nut OIT in young children. Once the first 12 participants have been enrolled, we will pause recruitment until all Pilot Phase participants in the Multi-Nut OIT Group have completed the build-up phase (~ 8 months). At this point we will undertake an interim analysis of the feasibility data, and review whether any adjustments need to be made to the protocol. Following this, and assuming that there are no major issues with the study protocol and further funding has been secured, we will continue recruitment into the trial as per the protocol.

Potential participants will be identified from these sources: public and private Allergy clinics, Centre for Food & Allergy Research (CFAR) and Allergy & Anaphylaxis Australia (A&AA) websites and social media. For the Pilot Phase, recruitment will begin with distribution of the 'LMNOP Study Invitation' flyer electronically via the CFAR website and email list (270+ families interested in participating in food allergy research), and on Facebook via the Murdoch Children's Research Institute (MCRI) and Melbourne Allergy Centre and Children's Specialists (MACCS) private allergy clinic. Parents who have expressed interest in the study will be contacted, and those children deemed likely to be eligible for the study according to study criteria following a screening phone call, will be invited to attend a 2-day screening assessment at the Melbourne Children's Trials Centre (MCTC), MCRI.

Screening day 1: Following informed parental consent, children will have a SPT and blood will be drawn. Children with a positive SPT (≥3mm) to 2 of peanut, cashew, almond, hazelnut or walnut will be offered 2 individual nut OFCs to confirm allergy and reaction thresholds prior to randomisation. The OFC will not be needed if the child's allergy history meets the study criteria for a confirmed allergy. The first OFC will take place on Screening day 1.

Screening day 2: Children will have a 2nd individual nut OFC. This will be completed approximately one week after the first OFC.

Once the child has completed screening and has confirmed IgE-mediated allergy to 2 peanut/tree nuts (positive SPT (≥3mm), and OFC), they will enter the treatment phase, and will be randomised to either:

Multi-Nut OIT Group: Participants will undergo multi-nut OIT treatment using a personalised multi-nut flour - 2 of peanut, almond, cashew, hazelnut or walnut, 1:1 ratio of allergen protein. Multi-Nut OIT Group participants will continue strict avoidance of confirmed allergens outside of their daily dose of multi-nut flour, and will have 24-hour access to an on-call study doctor in case of allergic reactions.

Standard Care Group: As per standard clinical care in Australia, families will be instructed to strictly avoid all confirmed nut allergens over the 18-month period.

The Multi-Nut OIT Group will undergo an 18-month treatment phase consisting of an escalation visit, build-up phase and maintenance phase as described above. Participants who pass their OFC after 18 months of OIT, and then another OFC after no OIT for 4 weeks for one or both of their study nuts, will enter the Ad libitum phase described above. After 12 months of this unrestricted consumption of the study nuts, with a minimum of approximately 300 mg protein per nut: ½ -1 teaspoon of nut flour, twice per week for both nuts, participants will be assessed for induced tolerance (IT) via another OFC. IT is when a child can eat standard serves of the food 12 months after stopping OIT, without having an allergic reaction.

The Standard Care Group for the 18 months will be instructed to avoid any consumption of the peanut/tree nuts they are allergic to, as per standard care. Participants who pass the OFC for one or both of their study nuts at the end of the 18 months will undergo the 12-month Ad libitum phase. At the end of this 12-month period, participants will then be assessed for maintaining NT via an OFC. That is, whether they have still outgrown their allergy.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 18 and 36 months at the time of Screening visit 1
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf
* IgE-mediated allergy to 2 of peanut, almond, cashew, hazelnut or walnut, confirmed by:

Nut 1 pre-screening:

For at least one of almond, cashew, hazelnut or walnut (Nut 1)*:

1. History of ingestion with IgE-mediated reaction (birth to present) AND
2. History of SPT ≥3mm OR History of sIgE ≥0.35 number of kilounits per liter (KuL) AND

Nut 2 pre-screening:

For a second nut out of peanut, almond, cashew, hazelnut or walnut (Nut 2):

History of SPT ≥3mm OR History sIgE ≥0.35 KuL

In clinic screening: Participants meeting pre-screening criteria for Nuts 1 and 2 above will be invited for in-clinic screening

1. SPT: wheal size ≥3mm at Visit 1 for 2 of peanut, almond, cashew, hazelnut or walnut AND
2. OFC: react to ≤3000 mg protein top dose (4449 mg cumulative) in open, single nut OFC for 2 of peanut, almond, cashew, hazelnut or walnut

OFC not needed if:

History of failed OFC within past 3 months (confirmed by investigator review of discharge summary) OR History of anaphylaxis after ingestion within past 3 months based on investigator judgement +/- review of ER/Ambulance/medical notes

*Peanut is not included as Nut 1 to reduce the incidence of screening children with a peanut allergy only - children with peanut allergy may have been advised to avoid all other nuts. We require children to have eaten and reacted to at least one tree nut, and then the 2nd nut, which children may or may not have eaten, can be peanut or a tree nut.

Exclusion Criteria:

* History of severe anaphylaxis (as defined by persistent hypotension, collapse, loss of consciousness, persistent hypoxia or ever needing more than 2 doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction)
* Severe anaphylaxis at study screening OFC (defined as persistent hypotension, collapse, loss of consciousness, persistent hypoxia, or requiring more than 2 doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction)
* Fails either screening OFC on dose 1 (0.5 mg).
* Underlying medical conditions that increase the risks associated with anaphylaxis (e.g., cardiac disease or poorly controlled asthma (defined below))
* Confirmed eosinophilic esophagitis (EoE) or history indicating EoE
* Current use of beta-blockers or angiotensin-converting enzyme (ACE) inhibitors
* Receiving systemic immunomodulatory treatment
* Not commenced or unable to eat solid food
* Weight <7.5kgs (recommended minimum weight for EpiPen Jr (adrenaline autoinjector))
* Has a sibling in the study

Defining uncontrolled asthma (Global Initiative for Asthma. Asthma management and prevention for adults and children older than 5 years)

In the past 4 weeks, has the patient had:

Daytime symptoms more than twice/week? Any night waking due to asthma? Short Acting Beta Agonist (SABA) reliever needed more than twice/week? Any activity limitation due to asthma? Uncontrolled - answered yes to 3-4 of these

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Main Trial: Comparison of the number of participants who pass their OFC after the 18-month treatment phase for both study nuts between the Multi-Nut OIT Group and Standard Care Group | At 18 months post commencement of treatment
  In both groups, passing requires participants tolerating all OFC doses for both of their study nuts. For the Multi-Nut OIT Group, participants must pass their OFC at the end of the 18-month treatment phase, and then pass another OFC after 4 weeks of no OIT. For the Standard Care Group, participants must pass their OFC after the 18-month period. Participants have a personalised combination of two nuts: a. peanut, b. almond, c. cashew, d. hazelnut, e. walnut, as nominated at study screening.

SECONDARY OUTCOMES:
Main Trial: Difference between the Multi-nut OIT Group in comparison to the Standard Care Group in the proportion and severity of reported adverse events (AE) related to study nut ingestion during the 18-month treatment phase | During the 18-month treatment phase
  Number and severity of AEs as assessed by standardised predetermined criteria, related to study peanut/tree nut ingestion from randomisation to end of the 18-month treatment phase collected via OFC and clinic visit observations and medical history taken, and parent questionnaire diaries.
Main Trial: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in mean change from screening to 18 months in quality of life scores for the children, measured by the Food Allergy Quality of Life-Parent Form (FAQL-PF) | Screening and at 18 months
  The Food Allergy Quality of Life Questionnaires (FAQLQ) are disease-specific health-related quality of life questionnaires for patients with food allergy. The FAQL-PF completed by parents of children aged 0-12 years, consists of 30 items over 3 domains: emotional impact, food anxiety, social and dietary restrictions. Total and domain scores are calculated by dividing the sum of completed items by the number of competed items.
Main Trial: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in mean change from screening to 18 months in quality of life scores for the parents using the ICEpop CAPability measure for Adults (ICECAP-A) | Screening and at 18 months
  The ICECAP-A questionnaire is a measure of capability well-being for adults. It has been developed in the United Kingdom (UK) using in-depth and semi-structured qualitative research with adults over the age of 18; values for the UK, obtained using best-worst scaling, are available. The instrument contains five attributes - stability, attachment, autonomy, achievement, and enjoyment, each with four levels. Research on the instrument's validity, reliability, feasibility of use and sensitivity to change are still ongoing.
Main Trial: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in mean change from screening to 18 months in State/Trait anxiety using the State/Trait Anxiety Inventory (STAI) | Screening and at 18 months
  The STAI is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Higher scores are positively correlated with higher levels of anxiety.
Main Trial: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in the number of allergy-related healthcare visits from randomisation to 18 months | Randomisation to 18 months
  Captured per number of hospitalisations, Emergency Room (ER) visits, physician office visits, and medications/number of prescriptions using linked data to Medicare healthcare usage (Medical Benefits Scheme (MBS) and Pharmaceutical Benefits Scheme (PBS)) and Victorian Data Linkage for hospital presentations (Victorian Admitted Episodes Dataset (VAED)).
Main Trial: Difference between the two groups in change in SPT wheal size at screening and at 18 months | Screening and at 18 months
  Measured by SPT wheal size for each child's study nuts at screening and at 18 months.
Main Trial: Difference between the two groups in change in levels of specific Immunoglobulin E (sIgE) at screening and at 18 months | Screening and at 18 months
  Measured by levels of sIgE for each child's study nuts at screening and at 18 months.
Main Trial: Difference between the two groups in change in levels of specific Immunoglobulin G4 (sIgG4) at screening and at 18 months | Screening and at 18 months
  Measured by levels of sIgG4 for each child's study nuts at screening and at 18 months.
Main Trial: Difference between the two groups in change in levels of component-resolved diagnostic (CRD) at screening and at 18 months | Screening and at 18 months
  Measured by levels of CRD for each child's study nuts at screening and at 18 months. CRD is an approach utilised to characterize the molecular components of each allergen involved in a sIgE-mediated response.
Main Trial: Difference between the two groups in change in levels of basophil activation test (BAT) at screening and at 18 months | Screening and at 18 months
  Measured by levels of BAT for each child's study nuts at screening and at 18 months.
Main Trial: Total number of missed doses overall (all participants) in the Multi-Nut OIT Group over the 18 month treatment phase | During the 18-month treatment phase
  Compliance will be measured by daily parent diary records of doses consumed. Total number of missed daily doses overall (all participants).
Main Trial: Mean number of missed daily doses per participant in the Multi-Nut OIT Group over the 18 month treatment phase | During the 18-month treatment phase
  Compliance will be measured by daily parent diary records of doses consumed. Total number of missed daily doses averaged per participant.
Main Trial Ad Libitum Phase: Comparison of the number of participants who pass their OFC after the 12 month Ad Libitum phase for both study nuts between the Multi-Nut OIT Group and Standard Care Group | At 32 months
  In both groups, passing requires tolerating all OFC doses for both of their study nuts.
Main Trial Ad Libitum Phase: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in the proportion and severity of reported AEs related to study nut ingestion during the 12-month Ad libitum phase | During the 12 month Ad libitum phase
  Number and severity of AEs as assessed by standardised predetermined criteria, related to study peanut/tree nut ingestion from the start to the end of the 12-month Ad libitum phase collected via end of trial OFC observation and medical history, and parent 1-monthly questionnaires.
Main Trial: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in mean change from the start to the end of the Ad libitum phase in quality of life scores for the children, measured by the FAQL-PF | At the 18-month treatment phase assessment and at the 12 month Ad libitum phase assessment
  The Food Allergy Quality of Life Questionnaires (FAQLQ) are disease-specific health-related quality of life questionnaires for patients with food allergy. The FAQL-PF completed by parents of children aged 0-12 years, consists of 30 items over 3 domains: emotional impact, food anxiety, social and dietary restrictions. Total and domain scores are calculated by dividing the sum of completed items by the number of competed items.
Main Trial Ad Libitum Phase: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in mean change from the start to the end of the Ad libitum phase in quality of life scores for the parents using the ICECAP-A | At the 18-month treatment phase assessment and at the 12 month Ad libitum phase assessment
  The ICECAP-A questionnaire is a measure of capability well-being for adults. It has been developed in the UK using in-depth and semi-structured qualitative research with adults over the age of 18; values for the UK, obtained using best-worst scaling, are available. The instrument contains five attributes - stability, attachment, autonomy, achievement, and enjoyment, each with four levels. Research on the instrument's validity, reliability, feasibility of use and sensitivity to change are still ongoing.
Main Trial Ad Libitum Phase: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in mean change from the start to the end of the Ad libitum phase in State/Trait anxiety using the STAI | At the 18-month treatment phase assessment and at the 12 month Ad libitum phase assessment
  The STAI is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Higher scores are positively correlated with higher levels of anxiety.
Main Trial Ad Libitum Phase: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in the number of allergy-related healthcare visits during the 12-month Ad libitum phase | During the 12-month Ad libitum phase
  Captured per number of hospitalisations, ER visits, physician office visits, and medications/number of prescriptions using linked data to Medicare healthcare usage (MBS/PBS) and Victorian Data Linkage for hospital presentations (VAED)
Main Trial Ad Libitum Phase: Difference between the two groups in change in SPT wheal size from 18-months treatment phase assessment to the 12-month Ad libitum phase assessment | At the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment
  Measured by SPT wheal size for each child's study nuts at the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment.
Main Trial Ad Libitum Phase: Difference between the two groups in change in levels of sIgE from 18-months treatment phase assessment to the 12-month Ad libitum phase assessment | At the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment
  Measured by levels of sIgE each child's study nuts at the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment.
Main Trial Ad Libitum Phase: Difference between the two groups in change in levels of sIgG4 from 18-months treatment phase assessment to the 12-month Ad libitum phase assessment | At the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment
  Measured by levels of sIgG4 for each child's study nuts at the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment.
Main Trial Ad Libitum Phase: Difference between the two groups in change levels of CRD from 18-months treatment phase assessment to the 12-month Ad libitum phase assessment | At the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment
  Measured by levels of CRD for each child's study nuts at the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment. CRD is an approach utilised to characterize the molecular components of each allergen involved in a sIgE-mediated response.
Main Trial Ad Libitum Phase: Difference between the two groups in change levels of BAT from 18-months treatment phase assessment to the 12-month Ad libitum phase assessment | At the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment
  Measured by levels of BAT for each child's study nuts at the 18-month treatment phase assessment and at the 12-month Ad libitum phase assessment.
Main Trial Ad Libitum Phase: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in the amount of study nut consumption during the Ad libitum phase | During the 12-month Ad libitum phase
  Amount of study nut consumption during the Ad libitum phase based on parent 1-monthly questionnaires.
Main Trial Ad Libitum Phase: Difference between the Multi-Nut OIT Group in comparison to the Standard Care Group in the frequency of study nut consumption during the Ad libitum phase | During the 12-month Ad libitum phase
  Frequency of study nut consumption during the Ad libitum phase based on parent 1-monthly questionnaires.
Pilot Phase: Number of children at screening who refuse, are eligible, or are ineligible | At study screening, up to 4 weeks before starting treatment
  Pilot Phase: At screening, number of children who:
  1. refuse to participate
  2. are eligible
  3. are ineligible (and reason)
Pilot Phase: Number of children at recruitment who agree or refuse to participate | At study recruitment, up to 4 weeks before starting treatment
  At recruitment, number of eligible children who:
  1. agree to be in the study
  2. who refuse to be in the study
Pilot Phase: Number of participants in the Multi-Nut OIT Group who complete escalation | At completion of first day of treatment
  Number of children in the Multi-Nut OIT Group who complete all escalation doses
Pilot Phase: Number of participants in the Multi-Nut OIT Group who complete the build-up phase | At completion of build-up, between 3-8 months after commencing treatment
  Number of participants in the Multi-Nut OIT Group who complete build-up
Pilot Phase: Number of participants in the Multi-Nut OIT Group and the Standard Care Group who withdraw, discontinue, and/or experience 1 or more protocol violations | During the 18 month treatment phase
  Number of participants in either arm who:
  1. withdraw
  2. discontinue the treatment prior to 18 months
  3. experience 1 or more protocol violations
Pilot Phase: Number and severity of AEs during the screening OFC for all participants | At study screening, up to 4 weeks before starting treatment
  Number and severity of AEs as assessed by standardised predetermined criteria during the screening OFC.
Pilot Phase: Number and severity of AEs for the Multi-Nut OIT Group during escalation | At completion of first day of treatment
  Number and severity of AEs as assessed by standardised predetermined criteria during escalation.
Pilot Phase: Number and severity of AEs for the Multi-Nut OIT Group during the build-up phase | During the build-up phase, between 3-8 month period after commencing treatment
  Number and severity of AEs as assessed by standardised predetermined criteria during build-up.
Pilot Phase: Total number of missed doses overall (all participants) in the Multi-Nut OIT Group over the build-up phase | During the build-up phase, between 3-8 month period after commencing treatment
  Based on parent diary entries. Number of missed daily doses overall (all participants).
Pilot Phase: Mean number of missed daily doses per participant in the Multi-Nut OIT Group over the build-up phase | During the build-up phase, between 3-8 month period after commencing treatment
  Based on parent diary entries. Number of missed daily doses averaged per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Perrett, MBBS FRACP, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set that will be collected for this analysis of the LMNOP trial will be available six months after publication of the primary outcome. The study protocol may be obtained from the Murdoch Children's Research Institute. Prior to releasing any data, the following are required: a data access agreement must be signed between relevant parties; the LMNOP trial investigators must see and approve the analysis plan describing how the data will be analysed; there must be an agreement around appropriate acknowledgment; and any additional costs involved must be covered.
  Should the study investigators be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognised research institute, which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months after the publication of the primary outcome
Access Criteria: Prior to releasing any data, the following are required: a data access agreement must be signed between relevant parties; the LMNOP trial investigators must see and approve the analysis plan describing how the data will be analysed; there must be an agreement around appropriate acknowledgment; and any additional costs involved must be covered.